CLINICAL TRIAL: NCT03212287
Title: Brilinta Tablets 60mg/90mg Clinical Experience Investigation
Brief Title: Brilinta Clinical Experience Investigation
Acronym: BRLCEIACS/OMI
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5133N00007
Record Dates: First submitted 2017-06-19; First posted 2017-07-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Acute Coronary Syndrome, Old Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
To confirm the following safety topics in patients to be treated with BRILINTA tablets 60 mg or 90 mg (hereinafter referred to as "BRILINTA") in clinical practice in the post-marketing phase.

1. Profile and incidence of ADRs The CEI will be conducted to collect data of the events, especially focusing on bleeding, dyspnoea and bradyarrhythmia so as to investigate onset, outcome, treatment for the event, and risk factors for these events, etc.
2. Profile and incidence of ADRs not expected from "Precautions for Use" of the ticagrelor JPI
3. Efficacy: Profile and incidence of cardiovascular events (cardiovascular death, non-fatal myocardial infarction and non-fatal ischemic stroke)
4. Factors which may affect safety or efficacy of ticagrelor

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with BRILINTA for ACS or OMI, which is the indication of the drug.

Exclusion Criteria:

-

Ages: 16 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with BRILINTA for ACS or OMI, which is the indication of the drug.
Sampling Method: Non-Probability Sample
Enrollment: 663 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | from baseline to 4 years
Incidence of ADRs not expected from "Precautions for Use" of the ticagrelor JPI | from baseline to 4 years
Incidence of cardiovascular events | from baseline to 4 years
Factors which may affect incidence of bleeding, dyspnoea, bradyarrhythmia, analysed by patient demographic characteristic and by treatment | from baseline to 4 years
Factors which may affect incidence of cardiovascular events, analysed by patient demographic characteristic and by treatment | from baseline to 4 years

CONTACTS AND LOCATIONS:
Locations (27):
- Japan (27):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Gunma
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Nagasaki
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokyo
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5133N00007&attachmentIdentifier=22799bd7-8c3b-461d-8da2-168b3d66eec9&fileName=Redacted_CSR_Synopsis_D5133N00007_Brilinta.pdf&versionIdentifier=